CLINICAL TRIAL: NCT02213055
Title: Safety and Efficacy of a 100% Dimethicone Pediculocide in School-Age Children
Brief Title: Pediatric Head Lice Study Product Comparison
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00000685
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Results first posted 2016-07-29 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-06

CONDITIONS: Head Lice
Keywords: Lice
MeSH Terms: conditions — Lice Infestations | interventions — Permethrin; Malathion; Hexachlorocyclohexane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LICEMD (Experimental): Infested children whose parents agree to use the investigational product will be enrolled on the experimental arm of the study using the LiceMD product as treatment.
  Interventions: Drug: LICEMD
- Standard Head lice product (Active Comparator): Parents/guardians who do not agree to use the investigational product and choose a standard head lice treatment will be asked to participate in the comparison arm of the study.
  Interventions: Drug: Standard Head lice product

INTERVENTIONS:
Drug: LICEMD — Parents/guardians of infested children will provide consent for their child's participation. Infested children whose parents agree to use the investigational product will be enrolled on the experimental arm of the study using the LiceMD product as treatment. Participants will be examined for lice count and scalp irritation the day after the first application, and one and two weeks after the first application.
  Other Names: Generic Name: Dimethicone
  Arms: LICEMD
Drug: Standard Head lice product — The most common treatments are pesticide-based, over-the-counter remedies of permethrin (1%), or pyrethrin-based products.After baseline scalp exam for lice count and preexisting signs of irritation, parents who agree to the comparison arm may purchase any other head lice treatment of their choice. All treatments are to be done at home by a parent or guardian. All participants will be examined for lice count and scalp irritation the day after the first application, and one and two weeks after the first application. Participants may also be examined by parents or the school nurse at any time if signs of irritation or re-infestation occur. If the child is still found to be infested during any examination, the school nurse will instruct the parent/guardian to retreat.
  Other Names: permethrin (5%); malathion (0.5%); lindane (1%)
  Arms: Standard Head lice product

SUMMARY:
* To evaluate the efficacy of LiceMD for the treatment of head lice in a pediatric population.
* To evaluate the safety of LiceMD in a pediatric population.

DETAILED DESCRIPTION:
Head lice, or Pediculus humanus capitis, cause an estimated 6 to 12 million infestations per year in the U.S., most commonly affecting children 3 to 11 years of age. Despite common perceptions, head lice crawl, and cannot hop or fly. For this reason, transmission occurs most often by human head-to-head contact, and much less commonly by the sharing of personal items such as hats, coats, combs, or towels. Because head lice feed on human blood, they cannot live on pets and are only viable 1-2 days on surfaces other than the human head.

ELIGIBILITY:
Inclusion Criteria:

* Subject Inclusion Criteria
* Current lice infestation, confirmed by school nurse. Must have live lice - not just eggs. A minimum of one live louse and 10 viable eggs must be seen or three live lice.
* Male or female child; age 3 - 12
* Willing to participate in study, and parent/guardian sign informed consent
* Parent/guardian must be able to read and follow directions and complete all questionnaires
* For children/parents who agree to the experimental arm of the study, agree not to use any other head lice product or home remedy lice treatment during the study.

Exclusion Criteria:

* No live lice, only eggs.
* Less than three live lice observed with less than ten viable eggs
* No hair on the head
* Buzz cut or crew cut
* Use of other lice treatment or home remedy lice treatment within the past 4 weeks
* Chronic scalp disorder (such as psoriasis) that would limit the school nurse's ability to detect lice and/or identify adverse events
* Currently taking an antibiotic
* Does not follow instructions.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2009-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Rosen, MD, Principal Investigator — Hackensack Meridian Health; Jeffrey Boscamp, MD, Study Director — Hackensack Meridian Health
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
The protocol and clinical dataset will be made available upon request to any scientist wishing to use them for non-commercial purposes.

REFERENCES:
- [Derived] Ihde ES, Boscamp JR, Loh JM, Rosen L. Safety and efficacy of a 100% dimethicone pediculocide in school-age children. BMC Pediatr. 2015 Jun 20;15:70. doi: 10.1186/s12887-015-0381-0. PMID 26092045

RESULTS

PARTICIPANT FLOW:
Groups:
- LICEMD: Infested children whose parents agree to use the investigational product will be enrolled on the experimental arm of the study using the LiceMD product as treatment.
  LICEMD: Parents/guardians of infested children will provide consent for their child's participation. Infested children whose parents agree to use the investigational product will be enrolled on the experimental arm of the study using the LiceMD product as treatment. All participants will be examined for lice count and scalp irritation the day after the first application, and at seven and fourteen days after the first application. Participants may also be examined by parents or the school nurse at any time if signs of irritation or re-infestation occur. If the child is still found to be infested during any of these examinations, the school nurse will instruct the parent/guardian to retreat.
- Standard Head Lice Product: Parents/guardians who do not agree to use the investigational product and choose a standard head lice treatment will be asked to participate in the comparison arm of the study.
  Standard Head lice product: The most common treatments are pesticide-based, over-the-counter remedies of permethrin (1%), or pyrethrin-based products. After a baseline scalp exam for lice count and preexisting signs of irritation, parents who agree to the comparison arm may choose and purchase any other head lice treatment of their choice. All treatments (investigational and comparison) are to be done at home by a parent or guardian. All participants will be examined for lice count and scalp irritation the day after the first application, and at seven and fourteen days after the first application.
Period: Overall Study
Arm/Group | LICEMD | Standard Head Lice Product
Started | 97 | 0
Completed | 58 | 0
Not Completed | 39 | 0
Not completed — Protocol was not Followed at Enrollment | 5 | 0
Not completed — Protocol was not Followed during Study | 1 | 0
Not completed — Documentation Issue at Enrollment | 1 | 0
Not completed — Documentation Issue during Study | 10 | 0
Not completed — Did not have Live Lice | 8 | 0
Not completed — Had another Treatment during the Study | 3 | 0
Not completed — Did not meet Inclusion Criteria | 6 | 0
Not completed — Did not Return to School | 5 | 0

BASELINE CHARACTERISTICS:
Population: There were 58 evaluable subjects in the experimental (LiceMD) arm of the study.
Groups:
- LiceMD: Infested children whose parents agree to use the investigational product will be enrolled on the experimental arm of the study using the LiceMD product as treatment.
  LiceMD: Parents/guardians of infested children will provide consent for their child's participation. Infested children whose parents agree to use the investigational product will be enrolled on the experimental arm of the study using the LiceMD product as treatment. All participants will be examined for lice count and scalp irritation the day after the first application, and at day seven and day fourteen after the first application. Participants may also be examined by parents or the school nurse at any time if signs of irritation or re-infestation occur. If the child is still found to be infested during any of these examinations, the school nurse will instruct the parent/guardian to retreat.
- Standard Head Lice Product: Parents/guardians who do not agree to use the investigational product and choose a standard head lice treatment will be asked to participate in the comparison arm of the study.
  Standard head lice product: The most common treatments are pesticide-based, over-the-counter remedies of permethrin (1%), or pyrethrin-based products. After a baseline scalp exam for lice count and preexisting signs of irritation, parents who agree to the comparison arm may choose and purchase any other head lice treatment of their choice. All treatments (investigational and comparison) are to be done at home by a parent or guardian. All participants will be examined for lice count and scalp irritation the day after the first application, and at day seven and day fourteen after the first application.
- Total: Total of all reporting groups
Arm/Group | LiceMD | Standard Head Lice Product | Total
Number analyzed (Participants) | 58 | 0 | 58
Age, Categorical [Number; unit: participants]
  <=18 years | 58 |  | 58
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 0 |  | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] — There were 58 evaluable subjects in the experimental (LiceMD) arm of the study.
  Years | 6.98 (1.73) |  | 6.98 (1.73)
Gender [Number; unit: participants]
  Female | 45 |  | 45
  Male | 13 |  | 13
Region of Enrollment [Number; unit: participants]
  United States | 58 |  | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Free of Live Head Lice and Free of Viable Eggs
Description: A determination of head lice effectiveness, measured by number of subjects free of live lice and by number of subjects free of viable eggs, was calculated using two week post-treatment data as the primary study outcome. Measurements were calculated at Day 1 (day after first treatment) and Day 14.
  At diagnosis, 55 subjects had viable eggs with three subjects meeting enrollment criteria for three or more live lice.
Time Frame: Day after first treatment and Day 14 of study
Population: There were 58 evaluable subjects in the experimental (LiceMD) arm of the study.
Measure: Number; unit: Participants
Groups:
- LiceMD: Infested children whose parents agree to use the investigational product will be enrolled on the experimental arm of the study using the LiceMD product as treatment.
  LICEMD: Parents/guardians of infested children will provide consent for their child's participation. Infested children whose parents agree to use the investigational product will be enrolled on the experimental arm of the study using the LiceMD product as treatment. All participants will be examined for lice count and scalp irritation the day after the first application, and at seven days and fourteen days after the first application. Participants may also be examined by parents or the school nurse at any time if signs of irritation or re-infestation occur. If the child is still found to be infested during any of these examinations, the school nurse will instruct the parent/guardian to retreat.
- Standard Head Lice Product: Parents/guardians who do not agree to use the investigational product and choose a standard head lice treatment will be asked to participate in the comparison arm of the study.
  Standard head lice product: The most common treatments are pesticide-based, over-the-counter remedies of permethrin (1%), or pyrethrin-based products. After a baseline scalp exam for lice count and preexisting signs of irritation, parents who agree to the comparison arm may choose and purchase any other head lice treatment of their choice. All treatments (investigational and comparison) are to be done at home by a parent or guardian. All participants will be examined for lice count and scalp irritation the day after the first application, and at seven days and fourteen days after the first application.
Arm/Group | LiceMD | Standard Head Lice Product
Number analyzed (Participants) | 58 | 0
Participants
  Day 1 Free of live lice | 57 |
  Day 14 Free of live lice | 55 |
  Day 1 Free of viable eggs | 32 |
  Day 14 Free of viable eggs | 46 |

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the period during which subjects were enrolled in the study, which was four years and one month.
Arm/Group | LiceMD | Standard Head Lice Product
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/0
Other Adverse Events (participants affected / at risk) | 1/97 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LiceMD (N=97) | Standard Head Lice Product (N=0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — School nurse transcribed adverse event (reported by parent/guardian), as "Irritation on cheek at time of shampoo application" which occurred "10 min after shampoo was washed off." Irritation lasted 10 minutes and no medical attention was needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No